CLINICAL TRIAL: NCT01401673
Title: Phase II Open-label Pilot Study of V3381, a Novel N-Methyl-D-Aspartate Receptor Antagonist, in Chronic Cough Patients Attending a Specialist Clinic
Brief Title: Phase II Open-Label Pilot Study of V3381 in Chronic Cough
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Vernalis (R&D) Ltd (Industry)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Development Director, Vernalis (R&D) Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V001
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Cough
Keywords: Chronic Cough; Indantadol
MeSH Terms: conditions — Cough; Chronic Cough | interventions — indantadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Indantadol — Titration

SUMMARY:
The investigators hypothesise that cough reflex hypersensitivity, demonstrated in chronic cough patients, is due to a phenomenon known as central sensitisation. Central sensitisation is a hyper-excitability of the sensory nerves as they join the central nervous system, and is believed to be mediated by the N-Methyl-D-Aspartate (NMDA) receptor[1-3].

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-75 years of age
* Females must be of non child-bearing potential
* Chronic Cough ( > 8 weeks)
* Normal Chest X-ray
* Normal Lung Function
* Idiopathic or treatment resistant cough-

Exclusion Criteria:

* Recent upper respiratory tract infection (<4 weeks)
* Pregnancy/breast-feeding
* Current smokers or ex-smokers with <6 months abstinence or cumulative history of >10 pack years
* Current treatment with ACE inhibitors.
* Drug or alcohol abuse
* Uncontrolled hypertension (i.e., >140/90 mmHg despite adequate medical therapy).
* Any cardiovascular condition that would be a contra-indication to the use of sympathomimetic amines (e.g. active angina).
* Any clinically significant neurological disorder
* Prior renal transplant, current renal dialysis.
* Any clinically significant or unstable medical or psychiatric condition that would interfere with the patient's ability to participate in the study.
* Increased risk of seizures.
* Any malignancy in the past 2 years (with the exception of basal cell carcinoma).
* Use of opioids, anticonvulsants, antidepressants (particularly MAO inhibitors).
* Any clinically significant abnormal laboratory test result(s).
* Serum creatinine laboratory value greater than 1.5 x upper limit of normal (ULN) reference range (after adjustment for age) or estimated creatinine clearance <60 mL/min.
* Total bilirubin greater than upper limit of normal reference range (with the exception of Gilbert's Syndrome) and/or alanine transaminase (ALT) >1.5 times upper limit of normal reference ranges (after adjustment for age).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Objective cough frequency at 8 weeks compared to baseline. | 8 Weeks

SECONDARY OUTCOMES:
Change in objective cough frequency at 4 weeks. | 4 Weeks
Change in Cough-Specific Quality-of-Life Questionnaire (CQLQ) at 4 and 8 weeks. | 4 and 8 Weeks
Change in Global Rating of Change Scale at 1 week, 2 weeks, 4 weeks and 8 weeks | 1 Week, 2 Weeks, 4 Weeks and 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Woodcock, Prof., Principal Investigator — South Manchester University Hospital
Locations (1):
- South Manchester University Hospital, Manchester, United Kingdom